CLINICAL TRIAL: NCT02317094
Title: Low-intensity Blood-flow Restricted Muscle Exercise in Patients With Sporadic Inclusion Body Myositis: a Randomised Controlled Trial
Brief Title: Blood-flow Restricted Exercise in Inclusion Body Myositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anders Nørkær Jørgensen, MSc. Sports Science, PhD student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20120166
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Sporadic Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Participants receive care as usual (various DMARDs, different from patient to patient).
  Interventions: Drug: Care as usual
- Blood-flow restricted tranining (Experimental): Participants will receive care as usual (various DMARDs, different from patient to patient) + 12 wks of low-intensity blood-flow restricted training twice per week.
  Interventions: Other: Blood-flow restricted training; Drug: Care as usual

INTERVENTIONS:
Other: Blood-flow restricted training — The intervention consists of low-intensity blood-flow restricted training involving 5 lower extremity exercises performed uni lateral in four sets to concentric failure with an intensity of approximately 25 repetition maximum (25RM).
  Arms: Blood-flow restricted tranining
Drug: Care as usual — The intervention consists of various DMARDs, which are given to the patients depending on their physical state and the disease activity.

SUMMARY:
This study evaluates the effects of a low-intensity blood-flow restricted exerciser protocol on patient reported physical function, in patients with sporadic inclusion body myositis. The study is designed as a parallel group randomized controlled trial with a treatment group and a control group.

DETAILED DESCRIPTION:
Sporadic inclusion body myositis (sIBM) is a disease characterized by skeletal muscle inflammation and severe muscle atrophy especially in the muscles in the thigh and the finger flexors. In time the muscle weakness will cause the affected person to become unable to walk and carry out basic tasks in the every day life.

Currently no effective treatment exist for sIBM patients, however several studies indicate that exercise may be beneficial for the patients.

In the resent years a lot of research attention has been directed toward low-intensity training with partial vascular occlusion as an alternative to the conventional high intensity strength training. Interestingly the low-intensity blood-flow occluded training is found to be at least as beneficial in causing muscle growth as the conventional strength training but with very little mechanical load on joints and tendons. Furthermore the blood-flow occluded training seem to result in a hyper-activation of muscle stem cells which play an important role in muscle regeneration.

This make the blood-flow restricted training modality a very interesting treatment possibility for sIBM patients because it might be able to restore and/or maintain the skeletal muscle tissue and therefore also muscle function.

ELIGIBILITY:
Inclusion Criteria:

Clinical features

* Duration of weakness > 12 months
* Weakness of finger flexors > shoulder abductors AND knee extension > hip flexion

Pathologic features

* Invasion of nonnecrotic fibres of mononuclear cells or rimmed vacuoles or
* increased major histocompatibility complex I (MHC-1) but no intracellular amyloid deposits or 15-18nm filaments

Exclusion Criteria:

* Lack of gait function
* Co-morbidity contraindicating the use of blood-flow restricted training (previous deep vein thrombosis/pulmonary embolism or known peripheral ischemic disease).
* Co-morbidity preventing resistance training (severe heart/lung-disease, uncontrolled hypertension (systolic > 160mmHg, diastolic > 100mmHg), severe knee/hip arthritis)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patient reported physical function (health survey (SF-36) subscale: Physical Function) | 12 wks
  Patient reported physical function will be evaluated with the short form (36) health survey (SF-36) subscale: Physical Function. The scale ranges from 0 to 100 where 100 is the highest score.

SECONDARY OUTCOMES:
Myositis Disease Activity Assessment Tool (MDAAT) | 12 wks
  An assessment tool used by the physician to evaluate disease activity in various organ systems via a scoring system and VAS scales.
Myositis Damage Index | 12 wks
  An assessment tool used by the physician to evaluate the damage caused by the disease or co-morbid conditions, to various organ systems. The system uses VAS scales.
Physician/Patient Global activity (VAS scale) | 12 wks
  A VAS scale used by both physician and patient to evaluate the overall activity of the disease
Physician/Patient Global Damage (VAS scale) | 12 wks
  A VAS scale used by both physician and patient to evaluate the overall damage caused by the disease.
2-min walk test | 12 wks
  A 2-min maximal walk test where the participant is encouraged to cover the greatest distance possible.
Manual Muscle Testing (MMT) | 12 wks
  A test of muscle strength in a series of muscles, carried out by the physician
Chair rise | 12 wks
  Participants are instructed to stand up and sit down on a chair as many times as possible in 30 sec.
Timed up & go | 12 wks
  Participants are instructed to rise from a chair walk 3 m forward, pass a marking and return to the chair and sit down as fast as possible
Health assessment questionnaire (HAQ) | 12 wks
  HAQ is a questionnaire to evaluate patient reported disability. It has 8 categories with a range of questions. Each question is scored from 0 to 3 where 0 is no disability and 3 is unable to do.
Inclusion body myositis functional rating scale (IBMFRS) | 12 wks
  A disease specific questionnaire evaluating the patients self reported everyday function.

OTHER OUTCOMES:
Blood samples | 12 wks
  Blood samples will be drawn for storage in a bio bank, for future analysis.
Muscle biopsies | 12 wks
  Muscle biopsies will be taken on a selected number of subjects from either the vastus lateralis or the tibialis anterior muscle, for the use in future analysis of i.e. muscle fibre size and distribution, myogenic stem cell activity, capillary density, muscle inflammation ect.
Sway - Postural Balance (using force plate) | 12 wks
  A test of postural balance
Maximal isometric and dynamic knee extension muscle strength (Kin-Com dynamometer) | 12 wks
  The maximal isometric and dynamic knee extension muscle strength will be evaluated in a Kin-Com dynamometer. Isometric strength data will be analyzed for peak torque, maximal impulse and maximal contractile rate of force development (RFD)
Leg extension muscle power (Nottingham Power Rig) | 12 wks
  The Nottingham Power Rig is used for evaluating the maximal muscle power that can be generated in the leg extensors.
Central activation (assessed with the twitch interpolation technique) | 12 wks
  Voluntary muscle activation will be assessed with the twitch interpolation technique.
Body composition ( full body duel energy X-ray absorption scan) | 12 wks
  Body composition will be evaluated with a full body duel energy X-ray absorption scan.

CONTACTS AND LOCATIONS:
Overall Officials: Anders N Jørgensen, PhD Student, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital (OUH), Odense, Fyn, Denmark

REFERENCES:
- [Background] Hilton-Jones D, Miller A, Parton M, Holton J, Sewry C, Hanna MG. Inclusion body myositis: MRC Centre for Neuromuscular Diseases, IBM workshop, London, 13 June 2008. Neuromuscul Disord. 2010 Feb;20(2):142-7. doi: 10.1016/j.nmd.2009.11.003. Epub 2010 Jan 13. No abstract available. PMID 20074951
- [Background] Alexanderson H. Exercise in inflammatory myopathies, including inclusion body myositis. Curr Rheumatol Rep. 2012 Jun;14(3):244-51. doi: 10.1007/s11926-012-0248-4. PMID 22467380
- [Background] Griggs RC, Askanas V, DiMauro S, Engel A, Karpati G, Mendell JR, Rowland LP. Inclusion body myositis and myopathies. Ann Neurol. 1995 Nov;38(5):705-13. doi: 10.1002/ana.410380504. No abstract available. PMID 7486861
- [Background] Era P, Heikkinen E. Postural sway during standing and unexpected disturbance of balance in random samples of men of different ages. J Gerontol. 1985 May;40(3):287-95. doi: 10.1093/geronj/40.3.287. PMID 3989241
- [Background] Bassey EJ, Short AH. A new method for measuring power output in a single leg extension: feasibility, reliability and validity. Eur J Appl Physiol Occup Physiol. 1990;60(5):385-90. doi: 10.1007/BF00713504. PMID 2369911
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] Aagaard P, Simonsen EB, Trolle M, Bangsbo J, Klausen K. Isokinetic hamstring/quadriceps strength ratio: influence from joint angular velocity, gravity correction and contraction mode. Acta Physiol Scand. 1995 Aug;154(4):421-7. doi: 10.1111/j.1748-1716.1995.tb09927.x. PMID 7484168
- [Background] Shield A, Zhou S. Assessing voluntary muscle activation with the twitch interpolation technique. Sports Med. 2004;34(4):253-67. doi: 10.2165/00007256-200434040-00005. PMID 15049717
- [Background] Lowes LP, Alfano L, Viollet L, Rosales XQ, Sahenk Z, Kaspar BK, Clark KR, Flanigan KM, Mendell JR, McDermott MP. Knee extensor strength exhibits potential to predict function in sporadic inclusion-body myositis. Muscle Nerve. 2012 Feb;45(2):163-8. doi: 10.1002/mus.22321. PMID 22246869
- [Result] Arnardottir S, Alexanderson H, Lundberg IE, Borg K. Sporadic inclusion body myositis: pilot study on the effects of a home exercise program on muscle function, histopathology and inflammatory reaction. J Rehabil Med. 2003 Jan;35(1):31-5. doi: 10.1080/16501970306110. PMID 12610846
- [Result] Spector SA, Lemmer JT, Koffman BM, Fleisher TA, Feuerstein IM, Hurley BF, Dalakas MC. Safety and efficacy of strength training in patients with sporadic inclusion body myositis. Muscle Nerve. 1997 Oct;20(10):1242-8. doi: 10.1002/(sici)1097-4598(199710)20:103.0.co;2-c. PMID 9324080
- [Result] Gualano B, Neves M Jr, Lima FR, Pinto AL, Laurentino G, Borges C, Baptista L, Artioli GG, Aoki MS, Moriscot A, Lancha AH Jr, Bonfa E, Ugrinowitsch C. Resistance training with vascular occlusion in inclusion body myositis: a case study. Med Sci Sports Exerc. 2010 Feb;42(2):250-4. doi: 10.1249/MSS.0b013e3181b18fb8. PMID 19927034
- [Result] Johnson, L.G., Edwards, D.J., Walters, S., Thickbroom, G.W., Mastaglia, F.L., The Effectiveness of an Individualized, Home-Based Functional Exercise Program for Patients With Sporadic Inclusion Body Myositis. J Clin Neuromuscul Dis 8(4): 187-194, 2007.
- [Derived] Jensen KY, Nielsen JL, Schroder HD, Jacobsen M, Boyle E, Jorgensen AN, Bech RD, Frandsen U, Aagaard P, Diederichsen LP. Lack of muscle stem cell proliferation and myocellular hypertrophy in sIBM patients following blood-flow restricted resistance training. Neuromuscul Disord. 2022 Jun;32(6):493-502. doi: 10.1016/j.nmd.2022.04.006. Epub 2022 Apr 26. PMID 35595645
- See also: Valuable knowledge about myositis diseases — http://www.myositis.org
- See also: Myositis evaluation tools — http://www.niehs.nih.gov/research/resources/imacs/othertools/index.cfm